CLINICAL TRIAL: NCT06795516
Title: Observational Study on the Clinical Use of ex Vivo Lung Perfusion (XPS™) for Lung Transplantation
Acronym: EVLP XPS
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: EVLP XPS 2023
Record Dates: First submitted 2025-01-17; First posted 2025-01-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-01

CONDITIONS: Lung Transplantation
Keywords: Ex-vivo Perfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Clinical use of ex-vivo perfusion for lung transplantation. Collection, storage and processing of patient data for outcome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Min Age 18 years
* Acceptance of the organ using the XPS™ ex vivo lung perfusion system is made by the center based on clinical assessment and visual inspection

Exclusion Criteria:

* The usual criteria for the assessment of donors apply
* The transplanting surgeon is not satisfied with the lung assessment on the XPS™ according to clinical criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Listed patients for lung transplantation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival of patients 1 year after transplantation | 1 year after transplantation

SECONDARY OUTCOMES:
Occurrence of primary graft dysfunction (PGD) after transplantation | 0, 24, 48, 72 hours postTx

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ius, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Department of Cardiothoracic, Transplant and Vascular Surgery, Hanover, Germany